CLINICAL TRIAL: NCT05145023
Title: Development and Validation of a Health-related Quality of Life Tool for Patients With Cardiac Sarcoidosis
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other); Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 143251; 256815 (Other: IRAS)
Record Dates: First submitted 2021-11-16; First posted 2021-12-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Sarcoidosis
Keywords: cardiac sarcoidosis; health-related quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Development of the CARD-SARC (n=20): * Interviews: 6-20 participants (depending of data saturation) will be recruited using a convenience sampling strategy.
  * Field-testing: 20 participants using a convenience/consecutive sampling strategy.
- Validation of the CARD-SARC (n=100): The CS-specialist centres (Barts Health NHS Trust and Royal Papworth Hospital NHS Foundation Trust) have a cohort of 60-70 potential candidates in each site. The estimated sample size for the Pilot-testing is 100 study participants, considering previous sarcoidosis studies including PROMs, with less than 10% population declining participation or failing to complete their questionnaires.

SUMMARY:
What is the purpose of this research?

This study includes two parts based in two NHS specialist centres for cardiac sarcoidosis:

* Development of the CARD-SARC: Development of the new questionnaire to measure quality of life in cardiac sarcoidosis patients (the CARD-SARC questionnaire)
* Validation of the CARD-SARC: Evaluation of how good the CARD-SARC questionnaire is at measuring quality of life changes in patients with cardiac sarcoidosis.

DETAILED DESCRIPTION:
What would taking part involve?

First, we would like to talk with a group of patients (between 6 to 20) about the impact of cardiac sarcoidosis in their quality of life during an interview. We will review and analysed these interviews. Then, we will compare with what is already know about cardiac sarcoidosis and its impact on quality of life. Also, we will ask healthcare professionals working with cardiac sarcoidosis patients to review our results. Finally, we will use this information to create the first draft of the new questionnaire (CARD-SARC questionnaire)to measure quality of life in cardiac sarcoidosis patients.

Second, we will ask 20 patients with cardiac sarcoidosis to complete the draft version of the CARD-SARC questionnaire. Also, they will complete validated quality of life questionnaires (for general population or sarcoidosis patients) and questionnaires that explore potential symptoms of fatigue, anxiety and depression. We will compare an review these results to confirm that the CARD-SARC questionnaire is ready for evaluation.

Third, we will ask 100 cardiac sarcoidosis patients to complete the CARD-SARC questionnaire and the validated questionnaires (for quality of life and potential sarcoidosis symptoms) to evaluate how good the CARD-SARC is at measuring quality of life changes in cardiac sarcoidosis patients.

How will patients or the public help guide the research?

This work has been influenced and designed with people living with cardiac sarcoidosis. SarcoidosisUK, the UK sarcoidosis charity, has been supportive and engaged on this work. Likewise, five expert patients with cardiac sarcoidosis have also agreed to lead, contribute and advice on relevant aspects of the study, and to participate sharing the results to the public, patients and professional groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years)
* Patients with a probable (50-90% likelihood) or highly probable (>90% likelihood) diagnosis of cardiac sarcoidosis (CS) by a multidisciplinary team meeting in a CS-specialist centre as per the WASOG criteria
* Patients attending outpatient clinics in a CS-specialist centre

Exclusion Criteria:

* Unable or unwilling to give informed consent
* Unable or unwilling to give and/or complete the study questionnaires • Inability to understand written and/or verbal English

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Using the WASOG criteria, participants will be adult patients attending the Outpatients Department with a probable (50-90% likelihood) or highly probable (>90% likelihood) diagnosis of cardiac sarcoidosis (CS) by a multidisciplinary team meeting in a CS-specialist centre.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To develop and validate a disease-specific HRQoL tool (CARD-SARC) for people diagnosed with cardiac sarcoidosis. | 12 months
  Patient-related research activities include semi-structured interviews for item generation (McMaster framework step 1 - item selection), field-testing for the development of the CARD-SARC questionnaire (McMaster framework step 3 - item reduction) and a pilot-testing for the validation of the CARD-SARC (steps 4-6 - determination of reliability, validity and responsiveness).

SECONDARY OUTCOMES:
The CARD-SARC questionnaire (new HRQoL-questionnaire for cardiac sarcoidosis). | 12 months
  To determine reliability, validity and responsiveness of the CARD-SARC:
  1. Internal consistency to determine if the CARD-SARC can be used as questionnaire to measure longitudinal changes in HRQoL in CS patients.
  2. Test-retest reliability to determine the concordance of two separated self-administration of the CARD-SARC.
  3. Longitudinal construct validity to determine the correlation between changes in the CARD-SARC and an external measure over time.
  4. Index of responsiveness for the CARD-SARC.
  The CARD-SARC will be self-completed by participants at baseline and weeks 2,12,24,52.
The 5-Levels of severity for the EuroQoL 5- Dimensions (EQ5D-5L) questionnaire. | 12 months
  This is a generic HRQoL/health status questionnaire. The EQ5D-5 consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each with five levels of health response and a visual analogue scale (VAS) ranging from 0-100 (0 being the worst possible health imaginable and 100 being the best possible health imaginable). The EQ5D-5L will be self-completed by participants at baseline and weeks 2,12,24,52 to assess HRQoL in CS patients using two standardised HRQoL-tools (EQ5D-5L and SF-36).
The Short-form 36 (SF-36) questionnaire. | 12 months
  This is a generic HRQoL/health status questionnaire. The SF-36 consists in eight scales eight dimension to measure two components: physical and mental summary scores ranging from 0-100. The physical component summary (PCS) includes physical functioning (10-items), role physical (4-items), bodily pain (2-items), general health (5-items). The mental component summary (MCS) includes vitality (4-items), social functioning (2-items), role emotional (3-items), mental health (5-items). Individual scores (0-100) can be obtained by weighted sums of the questions for each of the eight domains. The SF-36 will be self-completed by participants at baseline and weeks 2,12,24,52 to assess HRQoL in CS patients using two standardised HRQoL-tools (EQ5D-5L and SF-36).
The Sarcoidosis Health Questionnaire (SHQ) questionnaire. | 12 months
  This is a sarcoidosis-specific HRQoL questionnaire. The SHQ contains 29-items covering three domains: daily functioning, physical functioning, and emotional functioning. The responses range from "all of the time" (score of 1) to "none of the time" (score of 7). Higher score indicate better HRQoL. The SHQ will be self-completed by participants at baseline and weeks 2,12,24,52 to compare HRQoL in CS patients using three (non-cardiac) sarcoidosis-specific PROMs (SHQ, KSQ and SAT).
The King's Sarcoidosis Questionnaire (KSQ) questionnaire. | 12 months
  This is a sarcoidosis-specific HRQoL questionnaire. The KSQ contains 29-item covering five modules: general HRQoL (10- items), medications (3-items), lung (6-items), skin (3-items) and eyes (7- items). The KSQ is scored a re-ordered response scale ranging from 1 ("all of the time" or "a huge amount") to 7 ("none of the time" or "none at all"). The KSQ will be self-completed by participants at baseline and weeks 2,12,24,52 to compare HRQoL in CS patients using three (non-cardiac) sarcoidosis-specific PROMs (SHQ, KSQ and SAT).
The Sarcoidosis Assessment Tool (SAT). | 12 months
  This is a sarcoidosis-specific HRQoL questionnaire. The formatted version of the SAT contains 51-items covering components for physical functioning, satisfaction with roles and activities, fatigue, pain interference, sleep disturbance, sarcoidosis-lung concerns, sarcoidosis-skin concerns, and sarcoidosis-skin stigma. The responses ranging from 1 to 5 with different response options ("not at all" to "very much"; "unable to do" to "without any difficulty"; or "never" to "always"). The SAT will be self-completed by participants at baseline and weeks 2,12,24,52 to compare HRQoL in CS patients using three (non-cardiac) sarcoidosis-specific PROMs (SHQ, KSQ and SAT).
The Fatigue Assessment Scale (FAS). | 12 months
  The FAS is a one-dimensional fatigue questionnaire reflecting on physical (5-items) and mental fatigue (5-items). Each item has a five-point rating scare, ranging from "1-never" to "5-always". The score of FAS ranges from 10-50, with a well-defined cut-off for fatigue of >21 points. The FAS will be self-completed (optional) by participants at baseline and weeks 2,12,24,52 to assess fatigue in CS patients.
The Hospital Anxiety and Depression Scale (HADS). | 12 months
  The HADS is 14-item scale on a 4-point Likert scale (0-3) containing two subscales for anxiety and depression (7 items each subscale). The total score for each subscale is the sum of the respective items (ranging from 0-21). The HADS will be self-completed (optional) by participants at baseline and weeks 2,12,24,52 to assess anxiety and depression in CS patients.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - St Bartholomew's Hospital - Barts Health NHS Trust, London

IPD SHARING:
Plan to Share IPD: No